CLINICAL TRIAL: NCT03416023
Title: Prospective Multicentre Open Clinical Study to Assess the Safety Performance and Durability of the TIES® Transcutaneous Titanium Implant in Patients Requiring a Permanent Ileostomy
Brief Title: Safety, Performance and Durability of the TIES® Implant in Patients Requiring a Permanent Ileostomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The decision to halt the study is due to a discovered discrepancy between the study design and the anticipated use of the TIES product system.
  A new study will be launched during late 2024.
Sponsor: Ostomycure AB (Industry)
Collaborators: Devicia AB (now part of Veranex) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIES® III C03
Record Dates: First submitted 2018-01-10; First posted 2018-01-30 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Ileostomy - Stoma
Keywords: Implant; continence control; titanium

STUDY DESIGN:
Intervention Model Description: Prospective single-arm multicentre open clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single (Experimental)
  Interventions: Device: TIES® (Transcutaneous Implant Evacuation System)

INTERVENTIONS:
Device: TIES® (Transcutaneous Implant Evacuation System) — Transcutaneous Implant Evacuation System

SUMMARY:
Study to assess the safety, performance and durability of the TIES® transcutaneous titanium implant in patients requiring a permanent ileostomy.

DETAILED DESCRIPTION:
This is a multicentre, open-label, single-arm clinical study that will assess the safety, performance and durability of the TIES® transcutaneous titanium implant in patients requiring a permanent ileostomy (a surgical procedure that involves connecting the small intestine to the skin to create an opening).

The Transcutaneous Implant Evacuation System (TIES®) is a medical device designed to enable continence control for patients who would otherwise need to wear an ileostomy bag.

Eligible subjects will undergo a conventional ileostomy procedure under general anaesthesia and have the TIES® Port implanted. To date, the TIES® has been evaluated in 11 patients in 2 clinical studies. This study aims to collect more data that will assess performance, durability, safety and the impact that the TIES® has on a patient's quality of life.

The study will enroll 50 patients across Europe that require a permanent ileostomy, including patients with ulcerative colitis, familial adenomatous polyposis coli or other diseases such as Crohn´s disease.

Study subjects are expected to participate for approximately 1 year following surgical placement of the TIES® Port. Participation will involve a screening period, surgical implantation of the device (in-patient) and scheduled follow-up assessments out to 1 year post implant.

ELIGIBILITY:
Inclusion Criteria:

* Subject has ulcerative colitis, familial adenomatous polyposis coli or other diseases such as Crohn´s disease for whom a permanent ileostomy is indicated; or the subject has a medical need for an alternative to an existing conventional end-ileostomy, continent ileostomy or pelvic pouch; and
* Patient is a male ≥18 years of age or female ≥18 years of age (See exclusion criterion 4 regarding female with childbearing potential); and
* Signed written informed consent has been obtained prior to any study- related procedure.

Exclusion Criteria:

* Concurrent gastrointestinal fistula, parastomal or incisional hernia, or a history of recurrent gastrointestinal fistula, recurrent parastomal hernia(s), and/or recurrent incisional hernia(s).
* Patients with undetermined colitis.
* An acute episode of Crohn´s disease occurring during the last three months before the operation
* Females who are of childbearing potential and do not wish to use birth control measures for the duration of the study
* Patients receiving immunosuppressives, oncologic treatment or anticoagulants.
* Any clinically significant, abnormal, baseline laboratory result which in the opinion of the surgeon, affects the patient's suitability for the study or puts the patient at risk if he/she undergoes surgery
* Severe illness which, in the opinion of the surgeon may put the patient at risk when participating in the study or may affect the patient's ability to complete the study visits
* Condition associated with the risk of poor protocol compliance, e.g. alcoholism and/or drug abuse, dementia, self-destructive personality disorder
* Subjects with BMI ≤ 17 kg/m2 or BMI ≥ 33 kg/m2
* Participate in other clinical studies that could interfere with the result in the ongoing study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ludvig Linton, PhD, Study Director — OstomyCure AS
Locations (4):
- Sweden (2):
  - Gothenburgs University Hospital, Gothenburg
  - Linköpings University Hospital, Linköping
- United Kingdom (2):
  - St James' University Hospital, Leeds
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No
Currently no plan to share IPD but OstomyCure would be open to requests

RESULTS

PARTICIPANT FLOW:
Groups:
- TIES Implantation: TIES® (Transcutaneous Implant Evacuation System) implantation
Period: Overall Study
Arm/Group | TIES Implantation
Started | 28
Completed | 11
Not Completed | 17
Not completed — Exclusion criteria failure | 1
Not completed — Withdrawal by Subject | 6
Not completed — Explanted | 7
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Europe | 28

OUTCOME MEASURES:

1. Primary Outcome: Absence of Visible Leakage or Fecal Staining of Clothing at 24 Weeks
Description: Absence of visible leakage or fecal staining of clothing at 24 weeks after implantation of the TIES® Port.
Time Frame: 24 weeks after implantation of the TIES® Port
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 8
Participants | 2

2. Secondary Outcome: Absence of Visible Leakage or Fecal Staining of Clothing at 16 Weeks
Description: Absence of visible leakage or fecal staining of clothing at 16 weeks assessed in a diary
Time Frame: 16 weeks
Population: At 16 weeks
Measure: Number; unit: participants
Arm/Group | Single
Number analyzed (Participants) | 10
participants | 3

3. Secondary Outcome: Absence of Visible Leakage or Fecal Staining of Clothing 36 Weeks
Description: Absence of visible leakage or fecal staining of clothing at 36 weeks assessed in a diary
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 5
Participants | 2

4. Secondary Outcome: Absence of Visible Leakage or Fecal Staining of Clothing at 52 Weeks
Description: Absence of visible leakage or fecal staining of clothing at 52 weeks assessed in a diary
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Proportion of Implanted Subjects Using the TIES Lid at 16 Weeks
Description: Proportion of implanted subjects using the TIES Lid for continence control at 16 weeks
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 19
Participants | 10

6. Secondary Outcome: Proportion of Implanted Subjects Using the TIES Lid at 24 Weeks
Description: Proportion of implanted subjects using the TIES Lid for continence control at 24 weeks
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 19
Participants | 8

7. Secondary Outcome: Proportion of Implanted Subjects Using the TIES Lid at 36 Weeks
Description: Proportion of implanted subjects using the TIES Lid for continence control at 36 weeks
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 19
Participants | 5

8. Secondary Outcome: Proportion of Implanted Subjects Using the TIES Lid at 52 Weeks
Description: Proportion of implanted subjects using the TIES Lid for continence control at 52 weeks
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 19
Participants | 1

9. Secondary Outcome: Subject's Preferences Regarding Maintaining Body Hygiene
Description: Number of subjects who found it easier using the TIES® Lid than using stoma bags for periodic emptying of waste
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 8
Participants | 1

10. Secondary Outcome: Subject's Preferences Regarding Daily Activities
Description: Number of subjects who found it easier using the TIES® Lid than using stoma bags for periodic emptying of waste
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 8
Participants | 1

11. Secondary Outcome: Subject's Preferences: Being Worried About Odor From Stoma
Description: Number of subjects who were less worried when using the TIES® Lid than when using stoma bags for periodic emptying of waste
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 8
Participants | 1

12. Secondary Outcome: Subject's Preferences: Being Worried About Leakage From Stoma
Description: as for outcome 11
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 8
Participants | 1

13. Secondary Outcome: Subject's Preferences: Recommending the TIES Solution
Description: Number of subjects who would recommend the TIES solution to friends or family who need to undergo ileostomy
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single
Number analyzed (Participants) | 8
Participants | 1

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Single
All-Cause Mortality (participants affected / at risk) | 1/28
Serious Adverse Events (participants affected / at risk) | 9/28
Other Adverse Events (participants affected / at risk) | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=28)
Infection, implant site (Gastrointestinal disorders) | 1 (1)
Suspicion of pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1)
Self-explant of device (device misplacement or displacement) (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2)
Re-fashioning of ileostomy (Gastrointestinal disorders) | 1 (1)
Sepsis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (4)
Stenosis, stoma related event (Gastrointestinal disorders) | 1 (1)
Erythema at site (Skin and subcutaneous tissue disorders) | 1 (1)
Narrow passage caused by irritated or swollen intestine (Gastrointestinal disorders) | 2 (3)
Pain and redness following bowel resection to device (mucocutaneous separation/ peristomal skin lesi (Skin and subcutaneous tissue disorders) | 1 (1)
Infection and dehydration (Gastrointestinal disorders) | 1 (1)
Skin breakdown, pain, swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Dehiscence and leaking around the device (Gastrointestinal disorders) | 1 (1)
Pelvic infection (Gastrointestinal disorders) | 1 (2)
Incorrect ingrowth (Gastrointestinal disorders) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=28)
Cardiac event (Cardiac disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (5)
Granulation (Gastrointestinal disorders) | 1 (1)
Infection, blood (Blood and lymphatic system disorders) | 2 (4)
Infection, bowel (Gastrointestinal disorders) | 2 (3)
Infection, pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 4 (7)
Irritable bowel (Gastrointestinal disorders) | 4 (9)
Non-optimal ingrowth (Gastrointestinal disorders) | 4 (4)
Skin reaction (Skin and subcutaneous tissue disorders) | 11 (16)

LIMITATIONS AND CAVEATS:
The SARS-CoV-2 pandemic affected the recruitment rate, and the number of subjects who participated in and completed the investigation was few. Of those enrolled, there were many dropouts, e.g. due to leakage at the lid. The low number of evaluable study participants limited the assessment of the medical device performance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data need to be submitted by the PIs to the sponsor for review and comment at least 60 days prior to submission for publication, public dissemination, or review by a publication committee. All reasonable comments made by the sponsor shall be incorporated into the publication. The sponsor shall be entitled to make a reasoned request that publication be delayed for a period of up to 6 months from the date of first submission to the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT03416023/Prot_SAP_000.pdf